CLINICAL TRIAL: NCT04239612
Title: Fitforlife- a Study of Mentor Led Physical Exercise for Persons Affected by Psychosis
Brief Title: Fitforlife- Exercise in Care of Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Region Skåne (Unknown); Region Halland (Other)
Responsible Party: Principal Investigator, Yvonne Forsell, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102
Record Dates: First submitted 2019-10-28; First posted 2020-01-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Psychotic Disorders
Keywords: Psychotic disorders; Exercise; Cognition; Metabolic markers
MeSH Terms: conditions — Psychotic Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: All patients attending open care units for psychosis will be invited to participate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical exercise (Other): Specified circular training, 60 minutes, 1-3 times/week
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — Regular physical exercise in groups. Circular training: both strength and fitness

SUMMARY:
Persons affected by psychosis have a shorter life expectancy mainly due to metabolic disorders. This is partly due to the drugs but also to a sedentary life style.

It is often a life long disorder with decreased overall function and thus need of life long care, both informal and formal. It is also a highly stigmatising disorder.

We are aiming at adding peer mentor led regular physical exercise to the open care of psychosis. it is well-known that physical exercise increase overall function, decrease metabolic risk factors and increase cognition. By using educated peer mentors who will lead the exercise sessions this will have an anti-stigmatising effect and improve self-confidence.

DETAILED DESCRIPTION:
Purpose and aims The overall purpose is to integrate peer-mentor supervised regular physical exercise in the open care of persons affected by psychosis. For specific research questions see separate information.

Recruitment of units and mentors Psychiatric open care units who are responsible for care of persons affected by psychosis will be contacted. First in Stockholm then in the rest of Sweden.

Those who are interested will assign 1-2 local contact persons from the staff and recruit 4 potential peer mentors among their patients.

Peer mentor education The peer mentors will be educated to be able to lead physical exercise sessions for other patients. Two units (8 mentors) will be educated together and the local contact persons will also attend. The education consists of three half days and is lead by a person educated in health pedagogics and physical exercise. It consists of theory and practice about physical exercise sessions with focus on circular training. A lof of emphasis will be put put on leadership and encouragement. The curriculum of the education is based on the pilot study.

Recruitment of participants The local contact persons together with the health care staff at the local units will recruit participants to the exercise sessions.

They will also perform the initial and 6 month follow up examinations. In order to do this they will receive education and support from the research team. A carefully written instruction is administered. This procedure is described in detail in the study protocol.

Exercise sessions Each included unit will have exercise sessions at the unit. Numbers/week depends on the number of recruited participants. Schedule will be done by the local peer mentors and the local contact person together. The sessions will be entirely led by the peer mentors.

Before the sessions the local contact persons will register the participants when they arrive. After the session the peer mentor will report to the local contact person how the session went. These data will be transferred to the research team.

Support to the peer mentors For six months the educated peer mentors will have support from a health pedagogical team. The support is both face-to-face and electronic.

Time period The study will record data for 6 months.

ELIGIBILITY:
Inclusion Criteria:

• All persons attending open care psychiatric units for psychosis

Exclusion Criteria:

• Judged by the responsible psychiatrist that physical exercise in groups is not suitable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in overall function from baseline to 6 months | 6 months
  Overall function according to sum of items in WHODAS (World Health Organization Disability Assessment Schedule). 36 items, Score 0-5 on each item, higher values- lower function.

SECONDARY OUTCOMES:
Change in Body Mass Index(BMI) from baseline to 6 months | 6 months
  Weight and height will be combined to report BMI in kg/m2. Values >25 overweight, >30 obesity.
Change in Inflammatory markers from baseline to 6 months | 6 months
  Interleukin-6 (Il6), Tumour necrosis Factor (TNFalfa), C-reaktive protein(CRP) all measured in pg/ml. No normal values exists. Will be compared to healthy controls.
Changes from baseline to 6 months in cognitive function | 6 months
  Measured with Cogstate brief battery (Computerized congitive assessment) - score of the summarised tests. Generated through a computerized program, comparsion to age-matched controls.
Change in Glycated Hemoglobin (HBA1c ) | 6 months
  HBA1c measured in mmol/mol. Compared to normal values.
Change in fitness | 6 months
  Fitness measured as VO2 (Volyme Oxygene) max in a bicycle submax test (Ekblom-Bak). Will be compared to tables for normal values according to age.
Change in systolic and diastolic blood pressure | 6 months
  Blood pressure measured as mm hg. Will be compared to normal age related values.
Changes in blood lipids | 6 months
  Blood lipids includes cholesterol (LDL-C) measured in mg/dl, Low density lipoprotein (LDL) High density lipoprotein-cholesterol (HDL-C) and triglycerides- all measured in mg/dl. Will be compared to standard normal values according to age.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Forsell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm county council, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lambden B, Berge J, Forsell Y. Structured physical exercise and recovery from first episode psychosis in young adults, the FitForLife study. Psychiatry Res. 2018 Sep;267:346-353. doi: 10.1016/j.psychres.2018.06.001. Epub 2018 Jun 19. PMID 29957552
- [Result] Hallgren M, Skott M, Ekblom O, Firth J, Schembri A, Forsell Y. Exercise effects on cognitive functioning in young adults with first-episode psychosis: FitForLife. Psychol Med. 2019 Feb;49(3):431-439. doi: 10.1017/S0033291718001022. Epub 2018 May 6. PMID 29729687

DOCUMENTS (3):
  • Study Protocol (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04239612/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04239612/SAP_001.pdf
  • Informed Consent Form (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT04239612/ICF_002.pdf